CLINICAL TRIAL: NCT01711671
Title: A Pilot Study of DKN-01 and Lenalidomide (Revlimid®)/Dexamethasone Versus Lenalidomide/Dexamethasone in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: A Study of DKN-01 and Lenalidomide/Dexamethasone in Patients With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Leap Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DEK-DKK1-P101; DKN-01; LY2812176
Record Dates: First submitted 2012-10-18; First posted 2012-10-22 (Estimated); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Standard of Care; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- DKN-01 300mg (Experimental): DKN-01 plus lenalidomide (Revlimid)/dexamethasone
  Interventions: Drug: DKN-01 300 mg
- DKN-01 600mg (Experimental): DKN-01 plus lenalidomide (Revlimid)/dexamethasone
  Interventions: Drug: DKN-01 600 mg
- Standard of Care (Active Comparator): Lenalidomide (Revlimid)/dexamethasone
  Interventions: Drug: Standard of Care

INTERVENTIONS:
Drug: DKN-01 300 mg — 300 mg IV infusion of DKN-01 administered twice per 28 day cycle on Days 1 and 15, plus lenalidomide/dexamethasone
  Arms: DKN-01 300mg
Drug: DKN-01 600 mg — 600 mg IV infusion of DKN-01 administered twice per 28 day cycle on Days 1 and 15, plus lenalidomide/dexamethasone
  Arms: DKN-01 600mg
Drug: Standard of Care — Current approved standard of care
  Other Names: Lenalidomide; Revlimid; Dexamethasone
  Arms: Standard of Care

SUMMARY:
A study to evaluate the safety, efficacy and bone changes with combination therapy of intravenous (IV) infused DKN-01 and lenalidomide/dexamethasone, versus lenalidomide and dexamethasone in relapsed or refractory multiple myeloma (MM) patients

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory Multiple Myeloma (MM)

  a. Treated with at least 1 prior regimen for myeloma
  1. Prior treatment with bortezomib (Velcade) is acceptable with a wash-out of 2 weeks
  2. Treatment with prior autologous transplant is permitted
  3. If a transplant is used as consolidation following chemotherapy, without intervening disease progression, it will be considered 1 line of treatment with the preceding chemotherapy
* Diagnosis of symptomatic MM as defined by the International Myeloma Working Group (IMWG) :

  1. Second line or greater/Refractory/Relapsed, Stage I, Stage II, Stage III
  2. Measureable disease as indicated by monoclonal protein in the serum of greater than or equal to (≥) 1 grams per deciliter (g/dL), involved serum free light chain assay ≥10 mg/dL (≥100 mg/L) provided the serum free light chain ratio is abnormal; monoclonal light chain in the urine protein electrophoresis of ≥ 200 mg/24 hours, or measurable plasmacytoma
* At least 1 osteolytic bone lesion
* Disease-free of active second/secondary or prior malignancies for equal to or over 5 years with the exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in-situ" of the cervix or breast
* Ambulatory patients greater than or equal to (≥) 30 years of age
* Performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) scale
* Estimated life expectancy of ≥ 26 weeks
* Adequate organ function including:

  1. Hematologic:

     1. Absolute neutrophil count (ANC) greater than or equal to (≥) 1000/microliter
     2. Platelet (PLT) count ≥ 75,000/microliter
     3. Hemoglobin (Hgb) ≥ 8.0 g/dL
  2. Acceptable coagulation status:

     1. Prothrombin time (PT) and partial thromboplastin time (PTT) ≤ 1.2 x the upper limit of normal (ULN) unless receiving anticoagulation therapy. If receiving anticoagulation therapy, eligibility will be based upon International Normalization Ratio (INR)
     2. International normalized ratio (INR) less than or equal to (≤) 1.6 (unless receiving anticoagulation therapy)

        * If receiving warfarin: INR ≤ 3.0 (and no active bleeding, [i.e., no bleeding within 14 days prior to first dose of study therapy])
  3. Hepatic:

     1. Bilirubin ≤ 1.5 x ULN
     2. Alanine Transaminase (ALT) and Aspartate Transaminase (AST) ≤ 2.5 x ULN (if liver metastases are present, then ≤ 5 x ULN is allowed)
  4. Renal:

     1. Calculated creatinine clearance ≥ 45 mL using the Cockcroft and Gault Method
* Women of childbearing potential (WCBP) must have a negative serum or urine pregnancy test within 10 to 14 days and again within 24 hours of starting study drug

  1. WCBP must agree to have pregnancy tests monthly (every 14 days for women with irregular cycles) while on study drug and 4 weeks after the last dose of study drug
  2. Men must also agree to use a condom if their partner is of child bearing potential, even if they have had a successful vasectomy
  3. Males and females with reproductive potential must agree to use medically approved contraceptive precautions starting 4 weeks prior to initiation of the therapy and during the trial and for 18 months following the last dose of study drug
  4. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Provide written informed consent prior to any study-specific procedures
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures

Exclusion Criteria:

* Received treatment with an investigational drug, which has not received regulatory approval for any indication, within 28 days of study treatment with DKN-01
* Received any experimental non-drug therapy (e.g., donor leukocyte/mononuclear cell infusions) within 56 days of entry
* Previously treated with an anti-Dickkopf-1 (anti-DKK-1) or antibody therapy, or have had a significant allergy to a known pharmaceutical therapy that, in the opinion of the Investigator, poses an increased risk to the patient
* Received radiation therapy, surgery, or chemotherapy within 2 weeks prior to study entry (6 weeks for nitrosoureas or Mitomycin C)
* Received bisphosphonates (e.g., etidronate, clodronate, tiludronate, pamidronate, neridronate, olpadronate, alendronate, ibandronate, risedronate, zoledronate) within 2 weeks prior to study entry
* Symptomatic central nervous system (CNS) malignancy or metastasis. Patients with treated CNS metastases are eligible provided their disease is radiographically stable, asymptomatic, and they are not currently receiving corticosteroids and/or anticonvulsants. Screening of asymptomatic patients without a history of CNS metastases is not required
* Have a history of major organ transplant (for example: heart, lungs, liver, and kidney)
* Are pregnant or nursing
* Known to be human immunodeficiency virus (HIV) positive, have hepatitis B surface antigen (HBSAg), or hepatitis C antibodies (HCAb)
* Active, uncontrolled bacterial, viral, or fungal infections, including urinary tract infection, within 7 days of study entry requiring systemic therapy
* Serious cardiac condition such as myocardial infarction within the past 6 months, unstable angina, or Class III or IV congestive heart failure as defined by the New York Heart Association (NYHA); have ECG abnormalities including baseline 12-lead ECG with Fridericia-corrected QT interval (QTcF) > 470 msec (female) or > 450 msec (male), a history of congenital long QT syndrome, or any ECG abnormality that, in the opinion of the Investigator, would preclude safe participation in the study
* History of osteonecrosis of the hip or have evidence of structural bone abnormalities in the proximal femur on MRI scan that are considered clinically significant or may have an impact on the interpretation of the scan. Degenerative changes of the hip joint are not exclusionary
* Known concomitant disease(s) known to influence calcium metabolism including hyperparathyroidism, hyperthyroidism, Paget's disease of bone, or any other concurrent severe or uncontrolled concomitant medical condition that, in the opinion of the Investigator, would preclude participation in this study
* Patients who are currently receiving lithium chloride (LiCl)

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Fluorine F18 sodium fluoride positron emission tomography (NaF-PET/CT) standard uptake value (SUV) | Pre-study to after 6 months of therapy
  SUV as measured by NaF-PET/CT in both myeloma bone lesions and normal bone
Fluorine F18 sodium fluoride positron emission tomography (NaF-PET/CT) influx constant (Ki) | Pre-study to after 6 months of therapy
  Ki as measured by NaF-PET/CT in both myeloma bone lesions and normal bone
F18 fluorodeoxyglucose positron emission tomography (FDG-PET/CT) standard uptake value (SUV) | Pre-study to after 6 months of therapy
  SUV as measured by FDG-PET/CT in both myeloma bone lesions and normal bone
Number of patients with treatment emergent adverse events | Baseline to study completion (approximately 7 months)

SECONDARY OUTCOMES:
Overall response rate (ORR) | Baseline to study completion (approximately 7 months)
Progression free survival (PFS) | Baseline to study completion (approximately 7 months)
Duration of response | Baseline to study completion (approximately 7 months)
Overall survival | Baseline to study completion (approximately 7 months)
Pharmacokinetics: area under the concentration - time curve (AUC) of a single dose of DKN-01 | Dosing interval of 2 weeks following the first dose in Cycle 1
Pharmacokinetics: maximum plasma concentration (Cmax) of a single dose of DKN-01 | Dosing interval of 2 weeks following the first dose in Cycle 1
Pharmacokinetics: trough DKN-01 concentrations on Cycle 2 and Cycle 3 | Cycle 2 Day 1 Pre-dose, Cycle 3 Day 1 Pre-dose

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Sirard, Study Director — Leap Therapeutics
Locations (3):
- United States (3):
  - Emory University Hospital, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts